CLINICAL TRIAL: NCT03885583
Title: Evaluation of Post-operative Pulmonary Function After Open Kidney Surgery: Comparison Between Thoracic Epidural and Paravertebral Block
Brief Title: Post-operative Pulmonary Function After Kidney Surgery Under Two Different Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelbaky Abdelrahman, Assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: aunanesth202019
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Function
Keywords: kidney surgery; thoracic epidural block; paravertebral block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracic epidural group (Active Comparator): patients in this group will receive ultrasound guided thoracic epidural block preoperatively for pain management, continuous infusion of 0.5% bupivacaine through epidural catheter during operation and early post-operative period
  Interventions: Procedure: thoracic epidural block
- paravertebral group (Active Comparator): patients in this group will receive ultrasound guided pararvertebral block preoperatively for pain management, continuous infusion of paravertebral bupivacaine 0.5% through paravetebral catheter during operation and early post-operative period
  Interventions: Procedure: paravertebral block

INTERVENTIONS:
Procedure: thoracic epidural block — thoracic epidural block with bupivacaine 0.25% will be given in the 8th thoracic space using ultrasound
  Arms: thoracic epidural group
Procedure: paravertebral block — paravertebral block with 0.25 bupivacaine will be given at the level of the incision using ultrasound
  Arms: paravertebral group

SUMMARY:
To assess the respiratory and analgesic effects of continuous thoracic paravertebral block versus thoracic epidural in patients undergoing kidney surgery

DETAILED DESCRIPTION:
Study tools

* An Ultrasound machine (Madison X6) with superficial linear and curved probe.
* A 19 gauge echogenic needle and Plexolong Cather (PAJUNK, Plexolong Meier nanoline, Geisingen, Germany; 60 mm).
* A 17-gauge Tuohy needle and 19 G flex-tip catheter: for thoracic epidural.
* Spirometer: (Enraf-Nonius, Model SPIRO 601).
* Drugs: isobaric bupivacaine 0.25% (aside from the drugs used in the standard operation theatre).
* Computer software: computer generated random tables (for randomization) and SPSS 22 (for data analysis)

Thoracic epidural (TEP):

A pre-procedural ultrasound examination will be done to first identify the correct targeted thoracic level. To accomplish this, the transducer will be placed in the parasagittal plane approximately 5 cm from midline. The thoracic level will be determined by identifying the 12th rib and counting in a cephalad direction until the targeted level is marked.

All epidurals will be performed under all aseptic precautions with a 17-gauge Tuohy needle and 19 G flex-tip catheters. Using the loss of resistance to saline technique, catheters will be inserted 4 cm into the epidural space and a suitable test dose will be administered to exclude intravascular or sub-arachnoid injection

Bupivacaine 0.25% of 7.5-12 ml volume will be given through the epidural catheter then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15 ml/h with bolus infusion of 5 to 10 ml of the infusion mixture for breakthrough pain. The block height will be tested using pin prick method. After spirometry testing and diaphragmatic ultrasound, the infusion of TEP will be gradually weaned of and the catheter will be removed under complete aseptic precautions.

Thoracic paravertebral block: (TPVB) The Ultrasound-probe will be centered on T7. The sagittal technique at the transverse process, in-plane, will be used. The 19 gauge echogenic needle will be inserted in-plane at the lower border of the transducer and advanced in a cephalad position with real-time ultrasound sonography.

Injection of small amounts of fluid (hydro-dissection) will aid in needle tip location. When the needle tip reaches the paravertebral space, 7.5-12 ml Bupivacaine 0.25% will be slowly injected after negative aspiration. The endpoint for a successful block is anterior displacement of the pleura. The catheter will be then inserted through the needle and positioned up to 3 cm from skin entry directing upwards in the paravertebral space then continuous infusion of bupivacaine 0.1% will be infused at a rate of 5 ml/h up to 15 ml/h with bolus infusion of 5 to 10 ml of the infusion mixture for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA II, III
* elective kidney surgery

Exclusion Criteria:

* patient refusal
* contraindications to neuraxial blocks
* pneumonectomy
* planed postoperative mechanical ventilatoin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
vital capacity | 24 hours after operation
  measured by spirometer (Enraf-Nonius, Model SPIRO 601 medical Technologies)
forced vital capacity | 24 hours after operation
  measured by spirometer (Enraf-Nonius, Model SPIRO 601 medical Technologies)
forced expiratory volume in one second | 24 hours after operation
  measured by spirometer (Enraf-Nonius, Model SPIRO 601 medical Tecnologies)

SECONDARY OUTCOMES:
pain score | 24 hours after operation
  pain will be assessed using VAS score, it provides a range of scores from 0-100. A higher score indicates greater pain intensity.
diaphragmatic excursion | 24 hours after operation
  ultrasound assessment of diaphragmatic excursion

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed G Abdelraheem, MD, Study Director — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt